



## Cinnapoietin® Clinical Trial Protocol

A Phase III, randomized, two armed, multicenter, parallel, double blind (patient and assessor blinded), active controlled non inferiority clinical trial to determine the non-inferior therapeutic efficacy and safety between CinnaPoietin® (Beta erythropoietin) and Eprex® (epoetin alpha) on treatment of anemia in ESRD hemodialysis patients.

Date: 23 August 2015

NCT number: NCT03408639





## Cinnapoietin® clinical trial synopsis

| Title | A Phase III, randomized, two armed, multicenter, parallel, double blind (patient and assessor blinded), active controlled non inferiority clinical trial to determine the non-inferior therapeutic efficacy and safety between CinnaPoietin® (Beta erythropoietin) and Eprex® (epoetin alpha) on the treatment of anemia in ESRD hemodialysis patients |
|---|---|
| Aim of Study<br>(Primary objective) | Determination of non-inferior efficacy of Beta erythropoietin (CinnaPoietin®) compared with Eprex® (epoetin alpha) in correction of hemoglobin levels of anemic patients with chronic kidney disease (CKD) under hemodialysis |
| Secondary<br>objectives | The secondary outcomes of interest include assessment of efficacy and safety of Beta erythropoietin (CinnaPoietin®). |
| Study Design | The study is designed as phase III, randomized, two armed, multicenter, parallel, double blind (patient and assessor blinded), active controlled non inferiority clinical trial with primary outcome of hemoglobin level change in anemic patients with CKD under hemodialysis. |
| Registration | This study is planned to be registered in Iranian Registry of Clinical Trial (IRCT) |
| Sponsor | CinnaGen Co |
| Contract Research<br>Organization<br>(CRO) | CRO Trial, Tehran University of Medical Sciences, Tehran, Iran. |
| Principal<br>Investigator | Investigator name: Dr. Mohammad Reza Abbasi Affiliation: Nephrology Research Center, Tehran University of Medical Sciences, Tehran, Iran Recruitment centers: Ghiasi Hospital |





| Co-investigators<br>and recruitment<br>centers | 1. Dr. Jalal Azmandian Affiliation: Department of Nephrology, Kerman University of Medical Sciences, Kerman, Iran. Recruitment centers: 1. SHAFA Hospital 2. Javad Ol Aemeh Hospital 2. Dr Vahid Pourfarziani Affiliation: Nephrology and Urology Research Center, Baqyiatallah University of Medical Sciences, Tehran, Iran Recruitment centers: 1. Milad Hospital 3. Dr Shahrzad Ossareh Affiliation: Hasheminejad Kidney Center, Iran University of Medical Sciences, Tehran, Iran Recruitment centers: 1.Hashemi Nezhad Hospital 4. Dr Hooshang Sanadgol Affiliation: Hasheminejad Kidney Center, Iran University of Medical Sciences, Tehran, Iran Recruitment centers: 1. Hashemi Nezhad Hospital 5. Dr. Amirahmad Nasiri Affiliation: Imam Hossein Hospital, Shahid Beheshti University of Medical Sciences, Tehran, Iran Recruitment centers: 1. Imam Hossein Hospital 2. Madar Hospital 6. Dr Shahrokh Ezzat zadegan jahromi Affiliation: Nephro-Urology Research Center, Shiraz University of Medical Sciences, Shiraz, Iran Recruitment centers: 1. Haj Ebrahimi dialysis center |
|---|---|
| Investigational<br>Drug | Erythropietin beta biosimilar (CinnaGen co, Iran) |
| Comparator | Eprex® (erythropoietin alfa) (the reference drug, produced by Janssen-Cilag) |
| Sample size | 156 patients will be equally (1:1) divided into intervention arms (78 in each considering drop out) for achieving 80% power in order to determine non-inferiority using a one-sided, independent sample t-test. The margin of non-inferiority is -1. |





| | The true difference between the means is assumed to be -0.5. The |
|---|---|
| | significance level (alpha) of the test is 0.05. The data are drawn from populations with standard deviations of 1.2 and 1.2. |
| | Inclusion Criteria: |
| Eligibility criteria | <ul> <li>Inclusion Criteria:</li> <li>Aged between 18 and 70</li> <li>ESRD patients who are on hemodialysis for ≥3 months.</li> <li>Hb level 8-11.5 g/dl</li> <li>Patients are on adequate hemodialysis: the minimally adequate dose of hemodialysis given 3 times per week should be a spKt/V (single-pool delivered Kt/V; clearance of urea x dialysis time/volume of distribution) of 1.2 per dialysis. For treatment periods of less than 5 hours, an alternative minimum dose is a urea reduction rate (URR) of 65%. All types of hemodialysis systems and hemodiafiltration, including high-flux membranes are allowed as long as there is no plan to change the patient's regimen during the study.</li> <li>Sufficient iron stores, defined as serum ferritin ≥ 200 ng/ml and transferrin saturation ≥20%. (Patients not meeting these criteria may receive iron supplementation therapy during the Screening and stabilization period to appropriately correct their iron store deficiency to meet the criterion required for randomization);</li> <li>Ability to comply with study medication use, study visits, and study procedures as judged by the investigator;</li> <li>Females of childbearing potential agree to use an acceptable method of birth control (e.g., abstinence, hormonal or barrier methods, partner sterilization, or IUD) for the duration of the study.</li> <li>Qualified and willing to sign the informed consent form with the commitment of complying with all the scheduled visits, and study procedures as judged by the investigator;</li> <li>In any circumstances that potential participants are not able to give consent, it may be given by responsible parents or guardian.</li> <li>Exclusion criteria</li> <li>Uncontrolled hypertension (defined as pre-dialysis diastolic blood pressure ≥ 100 mmHg or systolic blood pressure ≥180 mmHg);</li> <li>Anemia secondary to other causes different to the CKD (e.g.</li> </ul> |
| | multiple myeloma, aplastic anemia, leukemia) |





- Decompensated liver failure;
- Clinical evidence of concurrent uncontrolled hyperparathyroidism (defined as serum parathyroid hormone (iPTH) > 800 pg/ml);
- Heart failure [New York Heart Association (NYHA) class III and IV];
- Unstable angina pectoris, active cardiac disease, stroke and/or cardiac infarction within the last six months;
- History of or active blood coagulation disorders including DVT, PTE, native access Thrombosis during last six months.
- Thrombocytosis (platelet count > 500,000/µl);
- Thrombocytopenia (platelet count < 100,000/µl);
- White blood cell count < 3,000/μl);
- White blood cell count  $> 15,000/\mu l$ )
- Recent Bleeding (acute or chronic bleeding within three months prior to screening);
- Suspicion of or confirmed occult bleeding (increased reticulocyte count);
- Clinical evidence of concurrent systemic infection, or inflammatory disease (e.g; diabetic foot, bed sore, access infection, CRP> 30 mg/l)
- Currently receiving treatment for epilepsy;
- Major surgery within 3 months prior to randomization and during the conduct of the trial (except vascular access surgery);
- Concomitant immunosuppressive therapy; patients on a short course of steroids (up to 7 days), topical or intranasal steroids are allowed in the study;
- History of any malignant disease within the last 5 years (except excised non-melanoma skin cancer);
- Women who are pregnant or breastfeeding;
- Known history of severe drug-related allergies;
- Known history of drug related allergy to Erythropoietin or one
  of the ingredients of the test or the reference products or
  hypersensitivity to mammalian-derived products;
- Transplant received within one year prior to the start of the study;





| | <ul> <li>Simultaneous participation in another clinical study or having received an Investigational Medicinal Product within three months before randomization in this study.</li> <li>Psychiatric, addictive (drugs or alcohol) or any other disorder that compromises the ability to give an informed consent;</li> <li>Any red blood cell transfusion during the last 3 months (measured at the time of eligibility verification);</li> <li>Primary hematological disorder (e.g. myelodysplastic syndrome, myeloma, sickle cell anemia, hematological malignancy, multiple myeloma hemolytic anemia);</li> <li>known resistance to the rHuEPO defined by a requirement &gt; 450 IU/kg/week by IV or 300 IU/kg/week by SC, equivalent to approximately 20.000 IU/week SC and in absence of iron deficiency;</li> <li>who have suffered an event of active bleeding in the 30 days prior to the beginning of the study;</li> <li>Morbid obesity, defined by a Body Mass Index (BMI) &gt; 37 kg/m2 in women and &gt; 40 kg/m2 in men.</li> </ul> |
|---|---|
| Pre Intervention | Pre-intervention treatment with iron will be of interest to reach a transferrin saturation percentage (TSAT) $\geq 20\%$ and a ferritin $\geq 200$ ng/ml. According to the KDIGO guidelines [41], if the TSAT is <20% and the serum ferritin <200 ng/ml (<200 µg/l) and an increase in Hb concentration without starting ESA treatment is desired, it is suggested to administer a trial of IV iron. IV iron may be provided as a single large dose or as repeated smaller doses depending on the specific IV iron preparation used (with the highest single dose varying by specific formulation). It is common practice to provide an initial course of IV iron amounting to approximately1000 mg; this may be repeated if an initial dose fails to increase Hb level and allow a decrease in ESA dose and if the TSAT remains <20% and serum ferritin remains <200 ng/ml (<200 mg/l) |
| Randomization | Cluster Randomization Method will be used to randomize patients in the study. The randomization monitor will create unblinding envelopes and packaged the drug with blinded labels. After the randomization, each patient will be given an identification code in order to be recognized |





| To prevent the influence of knowing interconclusion, the Subjects and those who a be unaware of the state of the patient with drugs or standard remedy. For this purpose, Subjects and administrusing a similar masked prefilled syringe identified by unique numbers. The treatment proposed in this study we KDIGO guidelines. Before the beginning to be able to enter the treatment, it shall stores are adequate. In addition to main /daily and B12 100 mcg (Amp)/monthly stores are adequates. Efficacy outcomes Primary outcomes: The mean Hb change level during The mean weekly epoetin dosage last 4 weeks of treatment neces within 10-12 g/dl during the last considered as a second primary entertains. | ator of drug will be blinded by es. All drugs packages will be as elaborated according to the of the protocol, for the patient be controlled that the iron (Fe) intervention, Nephrovit tablet |
|---|---|
| The treatment proposed in this study w KDIGO guidelines. Before the beginning to be able to enter the treatment, it shall stores are adequate. In addition to main /daily and B12 100 mcg (Amp)/monthly: Efficacy outcomes Primary outcomes: The mean Hb change level during The mean weekly epoetin dosage last 4 weeks of treatment neces within 10-12 g/dl during the last considered as a second primary en | of the protocol, for the patient<br>be controlled that the iron (Fe)<br>intervention, Nephrovit tablet |
| <ul> <li>Primary outcomes:</li> <li>The mean Hb change level during</li> <li>The mean weekly epoetin dosage last 4 weeks of treatment neces within 10-12 g/dl during the last considered as a second primary en</li> </ul> | |
| | per kg body weight during the sary to maintain the Hb level 4 weeks of treatment will be |
| <ul> <li>Secondary outcomes:</li> <li>The proportion of patients with an change during main study phase,</li> <li>The proportion of patients with an target range,</li> <li>Incidence of blood transfusions.</li> <li>Proportion of patients with treatm concentration≥11.0 g/dl AND two any blood transfusion within the part of mean Hb concentration of 11.0 consecutive weeks),</li> <li>Percentage of Hb measurements&gt;</li> </ul> | ent success (Hb consecutive weeks without |





| • | Percentage of hematocrit measurements>30% |
|---------------|-------------------------------------------|
| <u>Safety</u> | outcomes: |

- The incidence of Hb levels above 13 g/dL,
- Proportion of patients with an increase in Hb concentration of > 1.0 g/dL for 4 consecutive weeks,
- Incidence rate of adverse events

## **References:**

- 1. Astor, B.C., et al., Association of kidney function with anemia: the Third National Health and Nutrition Examination Survey (1988-1994). Archives of internal medicine, 2002. 162(12): p. 1401-1408.
- 2. Brittin, G., et al., Stability of blood in commonly used anticoagulants. Use of refrigerated blood for quality control of the Coulter Counter Model S. American journal of clinical pathology, 1969. 52(6): p. 690-694.
- 3. Locatelli, F., et al., Revised European best practice guidelines for the management of anaemia in patients with chronic renal failure. Nephrology, dialysis, transplantation: official publication of the European Dialysis and Transplant Association-European Renal Association, 2004. 19: p. ii1-47.
- 4. Wintrobe, M.M. and J.P. Greer, Wintrobe's clinical hematology. Vol. 1. 2009: Lippincott Williams & Wilkins.
- 5. Weiss, G. and L.T. Goodnough, Anemia of chronic disease. New England Journal of Medicine, 2005. 352(10): p. 1011-1023.
- 6. Fehr, T., et al., Interpretation of erythropoietin levels in patients with various degrees of renal insufficiency and anemia. Kidney international, 2004. 66(3): p. 1206-1211.
- 7. Rambod, M., C.P. Kovesdy, and K. Kalantar-Zadeh, Combined high serum ferritin and low iron saturation in hemodialysis patients: the role of inflammation. Clinical Journal of the American Society of Nephrology, 2008. 3(6): p. 1691-1701.
- 8. Aljama, P., et al., Serum ferritin concentration: A reliable guide to iron overload in uremic and hemodialyzed patients. Clinical nephrology, 1978. 10(3): p. 101-104.
- 9. Barany, P., et al., Serum ferritin and tissue iron in anemic dialysis patients. Mineral and electrolyte metabolism, 1996. 23(3-6): p. 273-276.
- 10. Blumberg, A.B., H.R.M. Marti, and C.G. Graber, Serum ferritin and bone marrow iron in patients undergoing continuous ambulatory peritoneal dialysis. JAMA, 1983. 250(24): p. 3317-3319.
- 11. Mirahmadi, K.S., et al., Serum ferritin level: determinant of iron requirement in hemodialysis patients. Jama, 1977. 238(7): p. 601-603.
- 12. Silverberg, D., et al., The effect of iv iron alone or in combination with low-dose erythropoietin in the rapid correction of anemia of chronic renal failure in the predialysis period. Clinical nephrology, 2001. 55(3): p. 212-219.





- 13. Fishbane, S., G.L. Frei, and J. Maesaka, Reduction in recombinant human erythropoietin doses by the use of chronic intravenous iron supplementation. American Journal of Kidney Diseases, 1995. 26(1): p. 41-46.
- 14. Sunder-Plassmann, G. and W. Hörl, Importance of iron supply for erythropoietin therapy. Nephrology Dialysis Transplantation, 1995. 10(11): p. 2070-2076.
- 15. Macdougall, I.C., et al., A randomized controlled study of iron supplementation in patients treated with erythropoietin. Kidney international, 1996. 50(5): p. 1694-1699.
- 16. Chang, C., C. Chang, and S. Chiang, Reduction in erythropoietin doses by the use of chronic intravenous iron supplementation in iron-replete hemodialysis patients. Clinical nephrology, 2002. 57(2): p. 136-141.
- 17. DeVita, M., et al., Targeting higher ferritin concentrations with intravenous iron dextran lowers erythropoietin requirement in hemodialysis patients. Clinical nephrology, 2003. 60(5): p. 335-340.
- 18. Navarro, J.F., et al., Effectiveness of intravenous administration of Fe-gluconate-Na complex to maintain adequate body iron stores in hemodialysis patients. American journal of nephrology, 1996. 16(4): p. 268-272.
- 19. Tessitore, N., et al., The role of iron status markers in predicting response to intravenous iron in haemodialysis patients on maintenance erythropoietin. Nephrology Dialysis Transplantation, 2001. 16(7): p. 1416-1423.
- 20. Rozen-Zvi, B., et al., Intravenous versus oral iron supplementation for the treatment of anemia in CKD: systematic review and meta-analysis. American Journal of Kidney Diseases, 2008. 52(5): p. 897-906.
- 21. Allegra, V., G. Mengozzi, and A. Vasile, Iron deficiency in maintenance hemodialysis patients: assessment of diagnosis criteria and of three different iron treatments. Nephron, 1991. 57(2): p. 175-182.
- 22. Palmer, S.C., et al., Meta-analysis: erythropoiesis-stimulating agents in patients with chronic kidney disease. Annals of internal medicine, 2010. 153(1): p. 23-33.
- 23. Pfeffer, M.A., et al., A trial of darbepoetin alfa in type 2 diabetes and chronic kidney disease. New England Journal of Medicine, 2009. 361(21): p. 2019-2032.
- 24. Parfrey, P.S. and T. Wish, Quality of life in CKD patients treated with erythropoiesis-stimulating agents. American Journal of Kidney Diseases, 2010. 55(3): p. 423-425.
- 25. Gandra, S.R., et al., Impact of erythropoiesis-stimulating agents on energy and physical function in nondialysis CKD patients with anemia: a systematic review. American Journal of Kidney Diseases, 2010. 55(3): p. 519-534.
- 26. Johansen, K.L., et al., Systematic review and meta-analysis of exercise tolerance and physical functioning in dialysis patients treated with erythropoiesis-stimulating agents. American Journal of Kidney Diseases, 2010. 55(3): p. 535-548.
- 27. Solomon, S.D., et al., Erythropoietic response and outcomes in kidney disease and type 2 diabetes. New England Journal of Medicine, 2010. 363(12): p. 1146-1155.
- 28. AHEMIÏ, K., KDIGO clinical practice guideline for anemia in chronic kidney disease. Kidney international, 2012. 2: p. 279.





## Participants timeline

| | Study Period | rudy Period | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening/ Intervention Allocation Post Allocation | | | | | | | | Close-<br>out | | |
| Time point | Visit0 | Visit 1 | Visit 2 | Visit3 | Visit4 | Visit5 | Visit6 | Visit7 | Visit8-1 | Visit8-2 | Visit9 |
| Day | -28 to 0 | 1 | 14<br>± 2 | 28<br>± 2 | 42<br>± 2 | 56<br>± 2 | 84<br>± 2 | 140<br>± 2 | 156<br>± 2 | 168<br>± 2 | 182<br>± 2 |
| Week | -4 - 0 | 0 | 2 | 4 | 6 | 8 | 12 | 20 | 22 | 24 | 26 |
| Screening | × | | | | | | | | | | |
| Informed consent | × | | | | | | | | | | |
| Allocation | × | | | | | | | | | | |
| Clinical evaluation. | × | × | × | × | × | × | × | × | × | × | × |
| Concomitant medication | × | × | × | × | × | × | × | × | × | × | × |
| Intervention | | × | × | × | × | × | × | × | × | × | |
| Adverse Event | | × | × | × | × | × | × | × | × | × | × |
| Drug accountability | | × | × | × | × | × | × | × | × | × | × |